CLINICAL TRIAL: NCT05267990
Title: Impact of a Coronary Artery Calcium-guided Primary Prevention of Major Coronary Heart Disease for Asymptomatic Coronary Artery Disease in Diabetes: a Prospective Cohort Study
Brief Title: Coronary Artery Calcium-guided Primary Prevention of Major Coronary Heart Disease in Asymptomatic Diabetes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: JuFeng, Hsiao (Other)
Collaborators: Lotung Poh-Ai Hospital (Other)
Responsible Party: Sponsor-Investigator, JuFeng, Hsiao, doctor, Lotung Poh-Ai Hospital
Organization: Lotung Poh-Ai Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB110-251-A
Record Dates: First submitted 2022-01-26; First posted 2022-03-07 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Type2 Diabetes; Coronary Heart Disease
Keywords: coronary artery calcium score; type 2 diabetes; coronary heart disease
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus, Type 2 | interventions — Multidetector Computed Tomography

STUDY DESIGN:
Intervention Model Description: a prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- coronary artery calcium-guide (Active Comparator): 1500 asymptomatic T2DM patients who will receive Coronary artery calcium (CAC) imaging using 256 sliced multi-detector computerized tomography (MDCT) scanner If CAC score >0, Treadmill ECG or Thallium201 Scan would be arranged. If Treadmill ECG or Thallium201 show significant ischemia, further study such as CT angiography or coronary angiography will be arranged.
  If CAC score > 100， Aspirin 100mg QD will be suggested to decrease the cardiovascular risk in patients with low risk of bleeding. Previous studies revealed aspirin for patients with CAC score>100 at low bleeding risk indicated net benefit If CAC score > 400，statin therapy will be suggested to control lipidemia aggressively and target LDL level<70 mg/dL
  Interventions: Diagnostic Test: Multi-Detector Computed Tomography
- usual care (No Intervention): The investigators will enroll 500 age, gender, risk factor matched T2DM patient from our hospital. The doctor in charge will give usual care according to the Diabetes associate of Taiwan clinical practice guidelines for diabetes care.

INTERVENTIONS:
Diagnostic Test: Multi-Detector Computed Tomography — Coronary angiography calcium score via Multi-Detector Computed Tomography
  Arms: coronary artery calcium-guide

SUMMARY:
To evaluate benefits of primary prevention of major coronary heart disease for asymptomatic coronary artery disease in type 2 diabetes mellitus based on the coronary artery calcium score Our proposal

1. Based on CAC score, primary early prevention could reduce incidence of major coronary heart disease (CHD) including cardiac mortality, acute myocardial infarction, coronary revascularization
2. based on CAC score, primary early prevention could reduce all cause mortality, cardiac mortality, cardiovascular disease, heart failure, ischemic stroke, heart failure associated hospitalization and chronic kidney disease and related clinical cost effect

DETAILED DESCRIPTION:
Background The patients with type two diabetes mellites increased gradually and heart disease and cerebral vascular disease is the fourth leading cause of mortality. According to the National Health Insurance Research Database (NHIRD) till 2014, incidence of coronary heart disease is 25.2% and heart failure is 3.77%。Multiple complication including chronic kidney disease and cerebrovascular diseases were also well-known.

A systematic review study of scientific evidence from across the world in 2007-2017 revealed cardiovascular disease (CVD) affected 32.2% overall; 29.1% had atherosclerosis, 21.2% had coronary heart disease (CAD), 14.9% heart failure, 14.6% angina, 10.0% myocardial infarction and 7.6% stroke. CVD representing 50.3% of all deaths is a major cause of mortality among people with type 2 Diabetes mellitus (T2DM) (1).A study in Asian population revealed patients with diabetes had a 1.89-fold risk of all-cause death and 2.0-fold risk of cardiovascular death compared with patients without diabetes(2) . However, most diabetes with CAD are asymptomatic.

Coronary artery calcium (CAC) score measured by multi-detector computerized tomography is a reliable measure of subclinical atherosclerosis. The presence, extent and progression of CAC have been shown to predict adverse cardiovascular events better than traditional risk factors and global risk scoring (3-7)。Our previous study in 2020 revealed CAC score could predict long-term cardiovascular outcomes in asymptomatic patients with T2DM (8). 2019 AHA/ACC Guideline on the Primary Prevention of Cardiovascular Disease and 2019 ESC/EAS Guidelines for the management of dyslipidaemias recommend CAC score as a decision making aid for personalized risk management in primary prevention (9,10).This prospective cohort study will invest the impact of a coronary artery calcium-guided primary prevention of major coronary heart disease for asymptomatic coronary artery disease in T2DM.

Objective To evaluate benefits of primary prevention of major coronary heart disease for asymptomatic coronary artery disease in T2DM based on the coronary artery calcium score Our proposal

1. Based on CAC score, primary early prevention could reduce incidence of major coronary heart disease (CHD) including cardiac mortality, acute myocardial infarction, coronary revascularization
2. based on CAC score, primary early prevention could reduce all cause mortality, cardiac mortality, cardiovascular disease, heart failure, ischemic stroke, heart failure associated hospitalization and chronic kidney disease and related clinical cost effect.

Method

Population:

The investigator will enroll 1500 asymptomatic T2DM patients who will receive Coronary artery calcium (CAC) imaging using 256 sliced multi-detector computerized tomography (MDCT) scanner as research group and 500 patients as control group from Lan-Yan Diabetes Shared Care Network (public health bureau, clinics, and regional hospital in Yilan County).

Inclusion criteria: more than 40 years old T2DM patients have any one cardiovascular risk as follows

1. total cholesterol>200mg/dl or low density lipoprotein (LDL) >100mg/dl
2. blood pressure>140/90mm/Hg or taking anti-hypertension agents
3. history of smoking
4. family history of early coronary heart diseases
5. proteinuria Exclusion criteria: history of cardiovascular diseases such as coronary heart disease, stroke, heart failure etc, pregnant

CAC Scores Measurement Coronary artery calcium (CAC) imaging was performed using an 256 sliced multi-detector computerized tomography (MDCT) scanner (Philips Brilliance 256) equipped with high-resolution detectors.

Intervention for study group Based on 2019 AHA/ACC Guideline on the Primary Prevention of Cardiovascular Disease and 2019 ESC/EAS Guidelines for the management of dyslipidemias and result of CAC score(9-12), the investigator will recommend the in-charged doctor to control the cardiovascular risk factors more aggressively. The study protocols are as follows If CAC score >0, Treadmill ECG or Thallium201 Scan would be arranged. If Treadmill ECG or Thallium201 show significant ischemia, further study such as CT angiography or coronary angiography will be arranged.

If CAC score > 100， Aspirin 100mg QD will be suggested to decrease the cardiovascular risk in patients with low risk of bleeding. Previous studies revealed aspirin for patients with CAC score>100 at low bleeding risk indicated net benefit ( If CAC score > 400，statin therapy will be suggested to control lipidemia aggressively and target LDL level<70 mg/dL The investigator will follow up these patients every 6 month, record their results of blood tests and medication for 5 years. Primary endpoint is major coronary heart disease including cardiac mortality, acute myocardial infarction, coronary revascularization. Second endpoint include all caused death, death due to cardiovascular disease, heart failure, stroke, admission for heart failure, chronic kidney disease and cost related to AMI, coronary heart disease, heart failure, stroke, chronic kidney disease etc.

Control group 500 age, gender, risk factor matched T2DM patients from our hospital will be enrolled. The doctor in charge will give usual care according to the Diabetes associate of Taiwan clinical practice guidelines for diabetes care.

ELIGIBILITY:
Inclusion Criteria:

more than 40 years old T2DM patients have any one cardiovascular risk as follows

1. total cholesterol>200mg/dl or low density lipoprotein (LDL) >100mg/dl
2. blood pressure>140/90mm/Hg or taking anti-hypertension agents
3. history of smoking
4. family history of early coronary heart diseases
5. proteinuria

Exclusion Criteria:

history of cardiovascular diseases such as coronary heart disease, stroke, heart failure etc, pregnant

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of major coronary heart disease | 5-year followup
  cardiac mortality, acute myocardial infarction and coronary revascularization

SECONDARY OUTCOMES:
rate of mortality | 5-year followup
  all caused death, death due to cardiovascular disease, heart failure and stroke
rate of admission | 5-year followup
  admission for heart failure, chronic kidney disease and stroke
medical expenditure | 5-year followup
  Medical expenditure, including both inpatient and outpatient costs, the total medical cost of index hospitalization due to Medical expenditure based on Taiwan National Health Insurance Research Database within 5 year- followup, including both outpatient costs and the total medical cost of hospitalization related to AMI, coronary heart disease, heart failure, stroke, chronic kidney disease

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Huan Lei, MD, Principal Investigator — cardiovascular center, Lo-Tung Poh-Ai Hospital, Taiwan
Locations (1):
- Lo-Tung Poh-Ai Hospital, Yilan, Taiwan

DOCUMENTS (2):
  • Study Protocol (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT05267990/Prot_000.pdf
  • Informed Consent Form (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT05267990/ICF_001.pdf